CLINICAL TRIAL: NCT01511614
Title: Identifying Neurobiological Mechanisms That Underlie Acute Nicotine Withdrawal and Drive Early Relapse in Smokers
Brief Title: Nicotine Withdrawal Symptoms and Smoking Relapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 999912474; 12-DA-N474
Record Dates: First submitted 2012-01-13; First posted 2012-01-18 (Estimated); Results first posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2023-07-25

CONDITIONS: Nicotine Dependence
Keywords: fMRI; tDCS
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Transcranial Direct Current Stimulation; Tobacco Use Cessation Devices; Varenicline; Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- active tDCS (Active Comparator): (1) anodal left-dlPFC + cathodal right-vmPFC stimulation, with anode over the left dlPFC and cathode over the right-vmPFC; (2) cathodal left-dlPFC + anodal right-vmPFC stimulation, in which polarity is reversed between the two electrodes
  Interventions: Device: Transcranial Direct Current Stimulation
- sham tDCS (Sham Comparator): To simulate the experience of tDCS stimulation, current is ramped on and turned off at the beginning and end of the tDCS session. An additional sham option is to have the current ramp up and down only at the beginning of the sham session, and not at the end. This second sham is supported in the literature as an effective blinding technique, which subjects cannot distinguish from active stimulation (Gandiga et al 2006, Brunoni et al 2012) . One of these sham options will be used for data that will be analyzed together, to be determined based on equipment capabilities and preliminary analysis of blinding efficacy in our cross over design. We will assess the efficacy of sham condition by providing participants and the investigator with a questionnaire on the MRI/tDCS session, wherein they will report whether they thought the tDCS session was active or sham. The MRI operator (or other non protocol personnel) will control active/sham conditions.
  Interventions: Device: sham
- Main Study - Treatment (Other): Healthy male and female adults who smokers are actively seeking treatment for smoking cessation were asked to complete three study phases: pre-treatment study visits, treatment visits and post-treatment follow-up visits.
  Pre-treatment (phase 1): 2 MRI sessions: dose-matched nicotine patch or placebo patch during a 36hr smoking abstinence period completed prior to each. Within ~ 2wks of their second scan visit, participants will have 1-3 pre-treatment preparation visits with a therapist.
  Treatment (Phase 2): 15-18 visits over ~16-19 weeks. First dose of varenicline (0.5 - 1mg/day), 1 week prior to their quit date followed by 12wks of daily varenicline (2mg/day) as well as weekly and biweekly 30min counseling sessions.
  Follow-up Phase 3: visits at 1, 6, and 12 months after their last treatment visit to assess quit status and smoking abstinence since last visit, complete a series of state measures and complete a 15-20 min scan session.
  Interventions: Drug: Nicotine patch; Drug: Placebo patch; Drug: Varenicline Pill; Drug: Placebo pill
- Main Study - Non-Treatment (Other): Healthy male and female adults who have a history of 1 or more years of consistently smoking cigarettes with a urine cotinine level corresponding to smoker status for the specific test being used, typically corresponding to a urine cotinine above about 200 ng/ml, but who are not currently seeking treatment for smoking cessation. Non-treatment seeking smokers will not set a quit date or make a quit attempt, will not complete a treatment program as part of this study and will not be followed up after they complete the two pre-treatment visits.
  Interventions: Drug: Nicotine patch; Drug: Placebo patch
- Main Study - Motivational Interviewing (Other): Current smokers who meet criteria for participation but who are not currently ready to enter treatment for smoking cessation. These subjects will receive motivational interviewing to prepare them for a tobacco cigarette quit attempt.
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Transcranial Direct Current Stimulation (tDCS), a type of Non-invasive Brain Stimulation (NIBS), has the potential to modify neuronal circuits by application of a subthreshold conductive current through the scalp. Two potential targets for tDCS as a smoking cessation aid are the dorsolateral pre-frontal cortex (dlPFC), a node of the ECN, and the ventromedial prefrontal cortex (vmPFC), a node of the DMN. tDCS can potentially strengthen the control of the ECN through excitatory stimulation of the dlPFC, and weaken the influence of the DMN (Lerman et al 2014) by inhibitory stimulation of the vmPFC. The tDCS model we will use is the neuroConn DC-Stimulator MR (neuroCare Group GmbH, Munchen, Germany).
  Arms: active tDCS
Device: sham — Sham Comparator
  Arms: sham tDCS
Drug: Nicotine patch — Dose-match Nicotine for non-deprived scan
  Arms: Main Study - Non-Treatment; Main Study - Treatment
Drug: Placebo patch — Nicotine deprived
  Arms: Main Study - Non-Treatment; Main Study - Treatment
Drug: Varenicline Pill — Treatment
  Arms: Main Study - Treatment
Drug: Placebo pill — Active comparator to varenicline
  Arms: Main Study - Treatment
Behavioral: Motivational Interviewing — Motivational Interviewing for smoking cessation preparation
  Arms: Main Study - Motivational Interviewing

SUMMARY:
Background:

- Smoking is thought to cause changes in the brain that lead to addiction and craving. Smokers who try to quit experience nicotine withdrawal symptoms that include irritability, anxiety, and difficulty concentrating. These symptoms make it difficult for people to stop smoking. Many people say that they continue smoking to help relieve these symptoms, often within the first week after trying to quit. Researchers want to study what is happening in the brain to cause these symptoms, which may help identify new ways to successfully quit smoking.

Objectives:

- To study nicotine withdrawal symptoms and brain function in smokers who stop smoking for 36 hours.

Eligibility:

- Individuals between 18 and 65 years of age who smoke at least 10 cigarettes per day. Participants must be able to stop smoking for 36 hours on two occasions.

Design:

Phase 1

* This study will involve three visits to the National Institute on Drug Abuse.
* NOT be able to smoke for 36 hours before the two imaging visits.
* Wear a nicotine skin patch or a placebo (fake) patch during your 36 hour smoking abstinence period and study visits.
* Have your blood drawn to test for levels of stress-related hormones.
* Complete multiple MRI scanning sessions that last about 1.5 to 2 hours each.
* Undergo EEG (brain waves) recording.
* Answer questionnaires about how you think and feel.
* Complete various tasks and procedures inside and outside of the MRI scanner.

Phase 2

* This study will involve thirteen visits to the National Institute on Drug Abuse.
* Set a quit date and develop a treatment plan with a study therapist.
* Take Chantix (varenicline) every day for a period of 12 weeks.
* Meet for weekly and biweekly counseling sessions with a therapist.
* Answer questionnaires about how you think and feel.

Phase 3

* This study will involve three visits to the National Institute on Drug Abuse.
* Complete an MRI scanning session that will last about 20min each visit
* Meet with a study staff member on each visit who will ask you questions about your smoking behavior and how you think and feel.

DETAILED DESCRIPTION:
Objective

The primary objective of the current protocol is to gain a greater understanding of the neurobiological mechanisms underlying acute nicotine withdrawal and contributing to the maintenance of, or return to smoking behavior among nicotine-dependent individuals, in the service of developing future smoking cessation treatments. The Nicotine Withdrawal Syndrome is a major cause of failed quit attempts in smokers, and targeting this time period for intervention may help improve smoking cessation outcomes.

Study Population

We will recruit treatment seeking and non-treatment seeking smokers, as well as matched non-smoker control participants.

Design

There are 3 arms included in this protocol, each of which aims to understand the neurobiology of the Nicotine Withdrawal Syndrome during the initial quit period, with the broader goal of increasing quit success rate in the future.

Main Study: To understand (1) the acute neurobiological effects of nicotine withdrawal on treatment-seeking and non-treatment seeking smokers, (2) the long term neurobiological outcomes of varenicline treatment and smoking cessation counseling at 1, 6, and 12 months. We will recruit 85 treatment seeking and 35 non-treatment seeking smokers for a within (nicotine deprivation), between (treatment-seeking status) subjects randomized, double blind, placebo controlled study.

Motivational Interviewing Arm: (1) To increase motivation and preparation for smoking cessation treatment among individuals who express an interest in quitting smoking but are not currently ready to enter treatment, in the service of increasing quit success rate and (2) to understand the neurobiological basis of motivation to quit smoking, and the interaction between motivation to quit and mechanisms that underlie acute nicotine withdrawal. We will recruit 300 current smokers interested in quitting smoking, but not yet ready to set a quit date.

Transcranial Direct Current Stimulation (tDCS) Arm: To understand the acute effect of tDCS on 3 large-scale brain networks dysregulated in nicotine addiction and withdrawal, the Default Mode Network, the Executive Control Network, and the Salience Network. We will enroll 60 non-treatment seeking smokers, with the expectation of 35 completers; and enroll 55 non-smoking controls, with the expectation of 45 completers, for a double blind, sham controlled, randomized crossover study. Smokers will be studied in nicotine abstinence and nicotine sated conditions, as in the Main Study design.

Outcome measures

Primary outcome measures:

1. Change in BOLD signal and FC related to task parameters, between drug (or tDCS) condition.
2. Behavioral performance on each of the tasks assessing inhibitory control processes, reward responsiveness, amygdala, striatal, BNST reactivity, impulsive decision making, cue reactivity and working memory (e.g., reaction time, error rate, hit rate, reward bias).
3. Self-reported craving, withdrawal symptoms and mood/affect
4. Smoking abstinence as determined by self-reported tobacco use, urine cotinine, and breath CO.

Secondary outcome measures:

1. MRS for glutamate concentration.
2. Plasma ACTH and cortisol.
3. Resting state CBF from ASL.
4. ERP and EEG measures.
5. Ratings and scores on self-report characterization measures.
6. Structural MRI and DTI data.
7. Resting state FC at 1, 6 and 12 months post-treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

All Subjects must:

* Be between the ages of 18-65.
* Be right-handed. Assessment tool(s): Edinburgh Handedness Inventory.
* Be in good health. Justification: Many illnesses may alter fMRI signals as well as cognitive processes and neural functioning. Assessment tool(s): Participants will provide a brief health history during phone screening, and undergo a medical history and physical examination with a qualified IRP clinician.
* Be free of current moderate to severe DSM-V Substance Use Disorder on any drug, except nicotine in smokers. Those with past moderate to severe use disorder on substances may be included, provided they are in sustained remission (and not on maintenance therapy for opioid use disorder) and are not intoxicated on the day of the imaging session. Justification: Moderate to severe use disorder on other substances may result in unique CNS deficits that could confound results and introduce excessive variance, while mild substance use disorder and substance use disorder in remission are common in community samples of smokers. Assessment tool(s): Computerized SCID or comparable assessment and DSM-5 substance use disorder assessment.
* Be able to abstain from alcohol and other recreational drugs for 24 hours before each imaging session, and able to moderate caffeine intake 12 hours before each imaging session. Justification: Recent substance use, including alcohol, and caffeine modulate neural functioning in a way that would complicate data interpretation. Assessment tool(s): Self-report, breathalyzer, and urine toxicology screen with follow up neuromotor assessment to ensure absence of acute impairment with positive urine test.
* Smokers must meet the additional criteria:

  * Have a urine cotinine level corresponding to smoker status for the specific test being used, typically corresponding to a urine cotinine above about 200 ng/ml, and have been smoking for at least 1 year. Justification: The present protocol is interested in neurobiological mechanisms that underlie nicotine withdrawal, and is thus contingent on the presence of nicotine dependence. Assessment tool(s): Selfreport, commercial urine cotinine test corresponding to smoker status for the specific test being used, typically corresponding to a urine cotinine above about 200 ng/ml.
  * Be able to abstain from smoking for 12 hours prior to MRI-tDCS study sessions. Justification: The present protocol will investigate the effect of acute nicotine withdrawal on cognitive processes and response to tDCS. Assessment: Self-report and expired CO levels
* In addition, non-smokers must meet:

  * Not have a history of daily cigarette smoking or have used any nicotine products continuously lasting more than a month, and no smoking or continuous use of any nicotine products within the past year. Assessment Tools: Self-report, urine cotinine test, and expired CO levels.

EXCLUSION CRITERIA:

All participants will be excluded if they:

* Are not suitable to undergo an fMRI experiment due to certain implanted devices (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips or other implanted metal parts), body morphology, or claustrophobia. Justification: MR scanning is one of the primary measurement tools used in the protocol. Assessment tool(s): Prospective participants will fill out an MRI screening questionnaire and undergo an interview with an MR technologist. Questions concerning suitability for scanning will be referred to the MR Medical Safety Officer. Prospective participants will be questioned about symptoms of claustrophobia and placed in the mock scanner during their first visit to assess for possible difficulty tolerating the confinement of the scanner and for ability to fit into the scanner.
* Have musculoskeletal abnormalities restricting an individual s ability to lie flat for extended periods of time. Justification: MR scanning sessions require participants to lie flat on their backs and remain perfectly still for approximately one hour. Therefore, conditions that would make that difficult (e.g. chronic back pain, significant scoliosis) will be exclusionary. Assessment tool(s): History and physical examination by a qualified IRP clinician, supplemented with a trial of lying in the mock scanner to assess comfort issues.
* Have HIV or Syphilis. Justification: HIV and Syphilis both can have central nervous system (CNS) sequelae, thus introducing unnecessary variability into the data. Assessment tool(s): Oral HIV followed by blood test if oral test is + and STS+ without adequate prior treatment
* Regularly or intermittently use any prescription (e.g., benzodiazepines, barbiturates), over-the-counter (e.g., cold medicine) medications that are likely to alter BOLD signal (neuronal-vascular coupling). Justification: The use of these substances may alter the fMRI signal and/or neural functions of interest in the current study. Assessment tool(s): History and comprehensive urine drug screening to detect benzodiazepines, antipsychotics, anticonvulsants, and barbiturates. Note: If a participant is intermittently taking a medication likely to affect BOLD signal, the participant may be excluded or if scanned, will be scanned in the same medication state for data continuity purposes (i.e. either all scan days are scheduled after 5 half-lives since last medication use; or all scan days are scheduled on medication).
* Have any current neurological illnesses including, but not limited to, seizure disorders, frequent migraines or on prophylaxis, multiple sclerosis, cerebrovascular accident, movement disorders (except essential tremor, so long as it would not interfere with study tasks such as button pressing), history of significant head trauma, or CNS tumor. Justification: Neurological diseases alter CNS function and, possibly, the neuronal-vascular coupling that forms the basis of the fMRI signal. Assessment tool(s): History and physical examination by a qualified IRP clinician, urine drug screening for anticonvulsants not disclosed by history. History of head trauma with loss of consciousness of more than 30 minutes or with post-concussive sequelae lasting more than two days, regardless of loss of consciousness, will be exclusionary. The MAI who will also retain discretion to exclude based on a history of neurological illness that may compromise data integrity.
* Have current major psychotic disorders, mania, substance-induced psychiatric disorders, or any current suicidal ideations or history of suicide attempts. Moderate to severe current symptoms of mood or anxiety disorders will be exclusionary as well. However, mild mood or anxiety disorder symptoms will not be exclusionary, whether medicated or unmedicated. The MAI will reserve the right to exclude on the basis of psychiatric history not explicitly described in this criterion. Justification: Psychiatric disorders involve the central neural system (CNS) and, therefore, can be expected to alter the fMRI measures being used in this study, however, some degree of mood and anxiety symptoms are common in community samples of smokers. Assessment tool(s): Computerized SCID or comparable assessment, and clinical interview confirmation by clinician.
* Are cognitively impaired or learning disabled. Justification: Cognitive impairment and learning disabilities may be associated with altered brain functioning in regions recruited during laboratory task performance. Cognitive impairment may affect one s ability to give informed consent. Assessment tool(s): History of placement in special-education classes as a consequence of serious learning problems and not solely as a consequence of behavioral problems, assessed during the History and Physical screening assessment.
* Have significant cardiovascular conditions that would make use of nicotine patch unsafe. Justification: Nicotine patch may cause significant arrhythmias in susceptible individuals. Assessment tool(s): History and physical exam, including 12-lead EKG.
* Have any other major medical condition, such as diabetes mellitus, that in the view of the investigators would compromise the safety of an individual during participation, or the quality of data obtainable. Justification: Many illnesses not explicitly covered here may increase risk or alter important outcome measures. Assessment tool(s): History and physical examination by a qualified IRP clinician and CBC, urinalysis, NIDA chemistry panel (liver function tests, electrolytes, kidney function). The following lab values will result in exclusion from the study:

  i. Hemoglobin < 10 g/dl

ii. White Blood Cell Count < 2400/microl

iii. Liver Function Tests > 3X upper limit of normal

iv. Serum glucose > 200 mg/dl

v. Urine protein > 2+

vi. Serum creatinine > 2 mg/dl

The MAI will retain discretion to exclude based on less extreme lab results. After the screening process has been completed, the MAI will take into account all data collected in order to decide if there is an existing medical illness that would compromise participation in this research.

* Are pregnant, planning to become pregnant, or breastfeeding. Females are instructed in the consent to use effective forms of birth control during the study period. Justification: study procedures and drugs used in the current protocol may complicate pregnancy or be transferred to nursing children. Assessment tool(s): Urine and/or serum pregnancy tests, and clinical interview. Urine pregnancy tests will be conducted at the beginning of each imaging visit.
* Are non-English speaking. Justification: To include non-English speakers, we would have to translate the consent and other study documents and hire and train bilingual staff, which would require resources that we do not have and could not justify given the small sample size for each experiment. Additionally, the data integrity of some of the cognitive tasks and standardized questionnaires used in this study would be compromised as they have only been validated in English. Most importantly, ongoing communication regarding safety procedures is necessary when participants are undergoing MRI procedures. The inability to effectively communicate MRI safety procedures in a language other than English could compromise the safety of non-English speaking participants. Assessment tool(s): self-report.

Treatment-seeking smokers will also be excluded if they:

* Have moderate to severe renal impairment. Justification. Given that renal secretion is varenicline s major route of clearance, kidney impairment may result in higher systemic levels of the drug than intended. Per Pfizer s chantix insert, varenicline pharmacokinetics were unchanged in subjects with mild renal impairment in comparison to those with normal renal function, whereas individuals with moderate and severe impairment presented with varenicline levels 1.5 and 2.1-fold higher, respectively. Assessment tool(s): Estimated glomerular filtration rate. Renal insufficiency with estimated creatinine clearance < 60 ml/min calculated by the Cockcroft-Gault equation will be excluded.
* Are diabetic. Justification. A recent case report describes multiple episodes of severe hypoglycemia experienced by a 51 year old Type-I diabetic after beginning varenicline treatment. The discontinuation of varenicline resolved any further hypoglycemic episodes. The safety of varenicline has not been investigated in patients with diabetes. Assessment tool(s): Casual plasma glucose testing. Individuals with glucose levels above 200 mg/dl may be further evaluated for diabetes using a fasting glucose test or be excluded.
* The following exclusion criteria are new for the tDCS study:

  * Participated in any brain stimulation session less than two weeks ago, or underwent brain stimulation exposure for treatment purposes in the last 6 months, including tDCS or transcranial magnetic stimulation (TMS). Justification: Prior exposure to brain stimulation may result in carry-over effects that could confound the results of this study. Participants may enroll in the study once the listed time periods have passed. Assessment tool(s): Participant medical history and physical (H&P).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2013-05-20 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Janes, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abulseoud OA, Ross TJ, Nam HW, Caparelli EC, Tennekoon M, Schleyer B, Castillo J, Fedota J, Gu H, Yang Y, Stein E. Short-term nicotine deprivation alters dorsal anterior cingulate glutamate concentration and concomitant cingulate-cortical functional connectivity. Neuropsychopharmacology. 2020 Oct;45(11):1920-1930. doi: 10.1038/s41386-020-0741-9. Epub 2020 Jun 19. PMID 32559759
- [Result] Aronson Fischell S, Ross TJ, Deng ZD, Salmeron BJ, Stein EA. Transcranial Direct Current Stimulation Applied to the Dorsolateral and Ventromedial Prefrontal Cortices in Smokers Modifies Cognitive Circuits Implicated in the Nicotine Withdrawal Syndrome. Biol Psychiatry Cogn Neurosci Neuroimaging. 2020 Apr;5(4):448-460. doi: 10.1016/j.bpsc.2019.12.020. Epub 2020 Jan 13. PMID 32151567

RESULTS

PARTICIPANT FLOW:
Groups:
- Main Study - Treatment: Healthy male and female adults who have a history of 1 or more of consistently years smoking cigarettes with a urine cotinine level corresponding to smoker status for the specific test being used, typically corresponding to a urine cotinine above about 200 ng/ml, and are actively seeking treatment for smoking cessation.
  Participants expected to a) complete the two pre-treatment scan visits; 2) set a quit date; 3) attempt to quit for at least 24 hours; 4) have their quit status established (i.e., relapsed vs abstinent) at 1, 6 and 12 months following their quit date.
- tDCS Arm - Smoker: Healthy nicotine-dependent adult participants who are current non-treatment seeking smokers
- tDCS - Non-Smoker; tDCS - Behavioral Pilot: Healthy non-smoking, non-drug dependent controls
Period: Overall Study
Arm/Group | Main Study - Treatment | Main Study - Non-Treatment | Main Study - Motivational Interviewing | tDCS Arm - Smoker | tDCS - Non-Smoker | tDCS - Behavioral Pilot
Started | 14 | 28 | 2 | 32 | 33 | 3
Completed | 3 | 19 | 2 | 19 | 30 | 3
Not Completed | 11 | 9 | 0 | 13 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Main Study - Treament: Healthy male and female adults who have a history of 1 or more of consistently years smoking cigarettes with a urine cotinine level corresponding to smoker status for the specific test being used, typically corresponding to a urine cotinine above about 200 ng/ml, and are actively seeking treatment for smoking cessation.
  Participants expected to a) complete the two pre-treatment scan visits; 2) set a quit date; 3) attempt to quit for at least 24 hours; 4) have their quit status established (i.e., relapsed vs abstinent) at 1, 6 and 12 months following their quit date.
- Main Study - Motivational Interviewing Arm: Current smokers who meet criteria for participation but who are not currently ready to enter treatment for smoking cessation. These subjects will receive motivational interviewing to prepare them for a tobacco cigarette quit attempt.
- Total: Total of all reporting groups
Arm/Group | Main Study - Treament | Main Study - Non-Treatment | Main Study - Motivational Interviewing Arm | tDCS Arm - Smoker | tDCS - Non-Smoker | tDCS - Behavioral Pilot | Total
Number analyzed (Participants) | 14 | 28 | 2 | 32 | 33 | 3 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 28 | 2 | 32 | 33 | 3 | 112
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 1 | 19 | 16 | 1 | 54
  Male | 6 | 19 | 1 | 13 | 17 | 2 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 2 | 0 | 4
  Not Hispanic or Latino | 14 | 27 | 2 | 31 | 31 | 3 | 108
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 10 | 17 | 2 | 14 | 18 | 1 | 62
  White | 3 | 11 | 0 | 14 | 11 | 1 | 40
  More than one race | 1 | 0 | 0 | 3 | 1 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 28 | 2 | 32 | 33 | 3 | 112

OUTCOME MEASURES:

1. Primary Outcome: BOLD Activation in Right ACC During Parametric Flanker Task tDCS Stimulation
Description: BOLD percent signal change in right Anterior Cingulate Cortex (rACC) during parametric flanker task. This table is during 2mA Anodal tDCS at the left Dorsolateral prefrontal cortex (dlPFC), 2mA Cathodal tDCS at left dlPFC, or sham stimulation (i.e. placebo). The 3 task conditions are congruent (i.e. flanker stimuli are identical to target) and medium and high levels of incongruent.
Time Frame: During tDCS or sham stimulation. Day 1 for non-smokers. Day 1 or 2 for smokers (counterbalanced for nicotine condidtion)
Measure: Mean (Standard Deviation); unit: Percent BOLD change
Groups:
- tDCS Arm - Non-smoker: Non-smokers scanned under 3 tDCS conditions: anodal-(L)dlPFC/cathodal-(R) vmPFC, reversed polarity, and sham.
- tDCS Arm - Sated Smoker: Nicotine cigarette smokers scanned under 3 tDCS conditions: anodal-(L)dlPFC/cathodal-(R) vmPFC, reversed polarity, and sham. Participants were 12 hours abstinent, but wearing a nicotine patch 2 hrs before the scan.
- tDCS Arm - Placebo Smoker: Nicotine cigarette smokers scanned under 3 tDCS conditions: anodal-(L)dlPFC/cathodal-(R) vmPFC, reversed polarity, and sham. Participants were 12 hours abstinent, but wearing a placebo patch 2 hrs before the scan.
Arm/Group | tDCS Arm - Non-smoker | tDCS Arm - Sated Smoker | tDCS Arm - Placebo Smoker
Number analyzed (Participants) | 28 | 15 | 15
Percent BOLD change
  Anodal left dlPFC stimulation, task congruent | 1.051567464 (0.613503334) | 0.867749333 (0.632271673) | 0.8973946 (0.764795369)
  Anodal left dlPFC stimulation, task medium incongruent | 1.143702607 (0.792691244) | 1.1765768 (0.707165736) | 1.0322936 (0.970342615)
  Anodal left dlPFC stimulation, task high incongruent | 1.338308679 (0.765383086) | 1.392077933 (0.818806467) | 1.154613533 (1.057797744)
  Cathodal left dlPFC stimulation, task congruent | 0.925731857 (0.73461226) | 0.863549133 (0.862738124) | 1.062994933 (0.992544203)
  Cathodal left dlPFC stimulation, task medium incongruent | 0.960205786 (0.738140954) | 0.986851467 (0.895053512) | 1.258576333 (1.087900913)
  Cathodal left dlPFC stimulation, task high incongruent | 1.161453536 (0.74433763) | 1.243763333 (0.985162535) | 1.451806467 (1.160555321)
  Sham stimulation, task congruent | 1.025226143 (0.527038736) | 0.6320986 (0.476573713) | 0.968123333 (0.691987432)
  Sham stimulation, task medium incongruent | 1.073017964 (0.700394341) | 0.800749733 (0.653128921) | 1.046178533 (0.907522718)
  Sham stimulation, task high incongruent | 1.35570925 (0.931955153) | 1.0759744 (0.717756041) | 1.251218733 (0.647266532)

2. Primary Outcome: dACC Glutamate
Description: Glutamate measured in the dorsal Anterior Cingulate Cortex (dACC) measured as a ratio to Creatine and Phosphocreatine. Cigarette smokers were 12 hour (overnight) abstinent, and had either a nicotine patch or a placebo patch placed 1-2 hours before scanning.
Time Frame: 12 hours nicotine abstinent (plus 1-2 hours after patch)
Population: Note that the treatment part of the main arm did not take place. As a consequence, all procedures performed were identical for both 'main arm - treatment' and 'main arm - non-treatment'. As these groups are thus identical, they are combined herein.
Measure: Mean (Standard Error); unit: ratio to Cr+PCr
Groups:
- Main Arm - Sated Smoker: Nicotine cigarette smokers. Participants were 12 hours abstinent, but wearing a nicotine patch starting 1-2 hours before the scan.
- Main Arm - Withdrawn Smoker: Nicotine cigarette smokers. Participants were 12 hours abstinent, and wearing a placebo patch starting 1-2 hours before the scan.
Arm/Group | Main Arm - Sated Smoker | Main Arm - Withdrawn Smoker
Number analyzed (Participants) | 30 | 30
ratio to Cr+PCr | 1.5 (.03) | 1.54 (.029)

3. Primary Outcome: Behavioral Accuracy on N-Back Working Memory Task
Description: Behavioral Performance on N-Back Working Memory Task. Task consisted of 0-back, 1-back and 3-back. In this task, participants respond with a button when the current stimulus is the same as the previous one (1-back), the one 3 stimuli earlier (3-back) or the letter 'D' (0-back) depending upon task condition. Table values are accuracy as a percentage (i.e total times they reponded correctly / total trials). This table is during 2mA Anodal tDCS at the left Dorsolateral prefrontal cortex (dlPFC), 2mA Cathodal tDCS at left dlPFC, or sham stimulation (i.e. placebo).
Time Frame: During tDCS or sham stimulation. Day 1 for non-smokers. Day 1 or 2 for smokers (counterbalanced for nicotine condition)
Measure: Mean (Standard Deviation); unit: Percent Correct
Groups:
- tDCS Arm - Withdrawn Smoker: Nicotine cigarette smokers scanned under 3 tDCS conditions: anodal-(L)dlPFC/cathodal-(R) vmPFC, reversed polarity, and sham. Participants were 12 hours abstinent, and wearing a placebo patch 2 hrs before the scan.
Arm/Group | tDCS Arm - Non-smoker | tDCS Arm - Sated Smoker | tDCS Arm - Withdrawn Smoker
Number analyzed (Participants) | 28 | 15 | 15
Percent Correct
  Percent Correct - Anodal left dlPFC stimulation, task Zero-Back Condition | 91.43 (15.11) | 97.56 (5.27) | 94.67 (5.75)
  Percent Correct - Anodal left dlPFC stimulation, task One-Back Condition | 89.88 (13.47) | 93.33 (10.84) | 87.11 (11.88)
  Percent Correct - Anodal left dlPFC stimulation, task Three-Back Condition | 58.93 (16.88) | 67.11 (18.89) | 58.89 (16.79)
  Percent Correct - Cathodal left dlPFC stimulation, task Zero-Back Condition | 94.40 (7.65) | 98.00 (3.74) | 85.11 (15.83)
  Percent Correct - Cathodal left dlPFC stimulation, task One-Back Condition | 89.40 (12.00) | 91.78 (9.83) | 80.22 (20.41)
  Percent Correct - Cathodal left dlPFC stimulation, task Three-Back Condition | 59.52 (14.28) | 69.78 (18.28) | 54.00 (15.18)
  Percent Correct - Sham stimulation, task Zero-Back Condition | 89.88 (21.27) | 94.89 (13.21) | 90.89 (10.80)
  Percent Correct - Sham stimulation, task One-Back Condition | 88.81 (16.81) | 94.00 (7.04) | 82.22 (17.31)
  Percent Correct - Sham stimulation, task Three-Back Condition | 60.36 (15.11) | 70.00 (16.86) | 57.56 (19.90)

4. Primary Outcome: Behavioral Reaction Speed on N-Back Working Memory Task
Description: Behavioral Performance on N-Back Working Memory Task. Task consisted of 0-back, 1-back and 3-back. In this task, participants respond with a button when the current stimulus is the same as the previous one (1-back), the one 3 stimuli earlier (3-back) or the letter 'D' (0-back) depending upon task condition. Table values are reaction time speeds. This table is during 2mA Anodal tDCS at the left Dorsolateral prefrontal cortex (dlPFC), 2mA Cathodal tDCS at left dlPFC, or sham stimulation (i.e. placebo).
Time Frame: During tDCS or sham stimulation. Day 1 for non-smokers. Day 1 or 2 for smokers (counterbalanced for nicotine condition)
Measure: Mean (Standard Deviation); unit: 1/sec
Arm/Group | tDCS Arm - Non-smoker | tDCS Arm - Sated Smoker | tDCS Arm - Withdrawn Smoker
Number analyzed (Participants) | 28 | 15 | 15
1/sec
  Reaction speed - Anodal left dlPFC stimulation, task Zero-Back Condition | 2.24 (.35) | 2.36 (.33) | 2.20 (.34)
  Reaction speed - Anodal left dlPFC stimulation, task One-Back Condition | 2.13 (.44) | 2.22 (.28) | 2.05 (.41)
  Reaction speed - Anodal left dlPFC stimulation, task Three-Back Condition | 1.91 (.59) | 1.78 (.44) | 1.64 (.49)
  Reaction speed - Cathodal left dlPFC stimulation, task Zero-Back Condition | 2.26 (.39) | 2.35 (.36) | 2.29 (.28)
  Reaction speed - Cathodal left dlPFC stimulation, task One-Back Condition | 2.16 (.51) | 2.28 (.36) | 2.07 (.36)
  Reaction speed - Cathodal left dlPFC stimulation, task Three-Back Condition | 1.85 (.63) | 1.82 (.41) | 1.62 (.39)
  Reaction speed - Sham stimulation, task Zero-Back Condition | 2.22 (.37) | 2.25 (.37) | 2.24 (.30)
  Reaction speed - Sham stimulation, task One-Back Condition | 2.11 (.52) | 2.17 (.42) | 2.04 (.40)
  Reaction speed - Sham stimulation, task Three-Back Condition | 1.84 (.55) | 1.82 (.45) | 1.71 (.52)

5. Primary Outcome: Behavioral Accuracy on the Parametric Flanker Task
Description: Behavioral Performance on Parametric Flanker Task. Task consisted of 3 levels of difficulty: congruent trials (where distractors are the same as the target; e.g. HHHHHHH), incongruent2 trials (where the 2 furthest distractors on each side were incongruent with the target; e.g. HHSSSHH) and incongruent3 trials (where all distractors are incongruent with the target; e.g. HHHSHHH). Table values are accuracy as a percentage (i.e total times they reponded correctly / total trials). This table is during 2mA Anodal tDCS at the left Dorsolateral prefrontal cortex (dlPFC), 2mA Cathodal tDCS at left dlPFC, or sham stimulation (i.e. placebo).
Time Frame: During tDCS or sham stimulation. Day 1 for non-smokers. Day 1 or 2 for smokers (counterbalanced for nicotine condition)
Measure: Mean (Standard Deviation); unit: Percent Correct
Arm/Group | tDCS Arm - Non-smoker | tDCS Arm - Sated Smoker | tDCS Arm - Withdrawn Smoker
Number analyzed (Participants) | 28 | 15 | 15
Percent Correct
  Percent Correct - Anodal left dlPFC stimulation, Congruent Condition | 98.87 (2.28) | 98.88 (1.59) | 98.83 (1.45)
  Percent Correct - Anodal left dlPFC stimulation, Incongruent2 Condition | 97.97 (3.80) | 98.50 (2.57) | 98.26 (3.11)
  Percent Correct - Anodal left dlPFC stimulation, Incongruent3 Condition | 93.62 (7.06) | 93.81 (7.75) | 89.89 (10.31)
  Percent Correct - Cathodal left dlPFC stimulation, Congruent Condition | 99.08 (1.56) | 98.88 (1.83) | 97.81 (1.86)
  Percent Correct - Cathodal left dlPFC stimulation, Incongruent2 Condition | 97.74 (4.00) | 99.04 (1.79) | 97.26 (3.74)
  Percent Correct - Cathodal left dlPFC stimulation, Incongruent3 Condition | 94.44 (5.15) | 92.72 (7.12) | 91.58 (9.16)
  Percent Correct - Sham stimulation, Congruent Condition | 98.88 (1.99) | 98.83 (3.05) | 98.57 (2.05)
  Percent Correct - Sham stimulation, Incongruent2 Condition | 98.08 (2.44) | 97.75 (4.17) | 96.95 (3.92)
  Percent Correct - Sham stimulation, Incongruent3 Condition | 94.42 (5.76) | 92.62 (6.96) | 90.83 (7.65)

6. Primary Outcome: Behavioral Reaction Speed on the Parametric Flanker Task
Description: Behavioral Reaction speed on Parametric Flanker Task. Task consisted of 3 levels of difficulty: congruent trials (where distractors are the same as the target; e.g. HHHHHHH), incongruent2 trials (where the 2 furthest distractors on each side were incongruent with the target; e.g. HHSSSHH) and incongruent3 trials (where all distractors are incongruent with the target; e.g. HHHSHHH). Table values are reaction time speeds. This table is during 2mA Anodal tDCS at the left Dorsolateral prefrontal cortex (dlPFC), 2mA Cathodal tDCS at left dlPFC, or sham stimulation (i.e. placebo).
Time Frame: During tDCS or sham stimulation. Day 1 for non-smokers. Day 1 or 2 for smokers (counterbalanced for nicotine condition)
Measure: Mean (Standard Deviation); unit: 1/sec
Arm/Group | tDCS Arm - Non-smoker | tDCS Arm - Sated Smoker | tDCS Arm - Withdrawn Smoker
Number analyzed (Participants) | 28 | 15 | 15
1/sec
  Reaction speed - Anodal left dlPFC stimulation- Congruent Condition | 2.31 (.26) | 2.37 (.29) | 2.23 (.23)
  Reaction speed - Anodal left dlPFC stimulation - Incongruent2 Condition | 2.17 (.24) | 2.21 (.26) | 2.08 (.22)
  Reaction speed - Anodal left dlPFC stimulation- Incongruent3 Condition | 1.94 (.21) | 1.95 (.22) | 1.90 (.14)
  Reaction speed - Cathodal left dlPFC stimulation- Congruent Condition | 2.33 (.27) | 2.40 (.31) | 2.25 (.24)
  Reaction speed - Cathodal left dlPFC stimulation- Incongruent2 Condition | 2.19 (.26) | 2.24 (.28) | 2.13 (.27)
  Reaction speed - Cathodal left dlPFC stimulation- Incongruent3 Condition | 1.97 (.26) | 1.99 (.21) | 1.94 (.17)
  Reaction speed - Sham stimulation - Congruent Condition | 2.37 (.29) | 2.36 (.30) | 2.24 (.24)
  Reaction speed - Sham stimulation- Incongruent2 Condition | 2.19 (.27) | 2.18 (.26) | 2.11 (.26)
  Reaction speed - Sham stimulation- Incongruent3 Condition | 1.98 (.26) | 1.95 (.20) | 1.90 (.18)

7. Primary Outcome: Behavioral Accuracy on the Matching Task
Description: Behavioral Performance on the Matching Task. Task consisted of 2 conditions: match faces, where 2 faces appeared at the top of the screen and one at the bottom (target). Participants needed to press a button corresponding to the top row face that matched the target; the control condition was identical, except instead of faces the images consisted of simple shapes (e.g. ovals). Table values are accuracy as a percentage (i.e total times they reponded correctly / total trials). This table is during 2mA Anodal tDCS at the left Dorsolateral prefrontal cortex (dlPFC), 2mA Cathodal tDCS at left dlPFC, or sham stimulation (i.e. placebo).
Time Frame: During tDCS or sham stimulation. Day 1 for non-smokers. Day 1 or 2 for smokers (counterbalanced for nicotine condition)
Measure: Mean (Standard Deviation); unit: Percent Correct
Arm/Group | tDCS Arm - Non-smoker | tDCS Arm - Sated Smoker | tDCS Arm - Withdrawn Smoker
Number analyzed (Participants) | 28 | 15 | 15
Percent Correct
  Percent Correct - Anodal left dlPFC stimulation, shapes condition | 96.09 (4.14) | 98.33 (2.17) | 96.58 (4.80)
  Percent Correct - Anodal left dlPFC stimulation, faces condition | 98.28 (2.22) | 97.02 (3.81) | 96.08 (3.64)
  Percent Correct - Cathodal left dlPFC stimulation, shapes condition | 97.84 (3.17) | 97.36 (4.19) | 97.11 (4.89)
  Percent Correct - Cathodal left dlPFC stimulation, faces condition | 97.08 (3.85) | 96.43 (5.13) | 93.84 (7.77)
  Percent Correct - sham stimulation, shapes condition | 96.28 (4.43) | 97.86 (2.11) | 95.29 (6.54)
  Percent Correct - sham stimulation, faces condition | 98.21 (3.09) | 97.92 (3.56) | 94.70 (4.34)

8. Primary Outcome: Behavioral Reaction Speed on the Matching Task
Description: Behavioral Reaction speed on the Matching Task. Task consisted of 2 conditions: match faces, where 2 faces appeared at the top of the screen and one at the bottom (target). Participants needed to press a button corresponding to the top row face that matched the target; the control condition was identical, except instead of faces the images consisted of simple shapes (e.g. ovals).Table values are reaction time speeds. This table is during 2mA Anodal tDCS at the left Dorsolateral prefrontal cortex (dlPFC), 2mA Cathodal tDCS at left dlPFC, or sham stimulation (i.e. placebo).
Time Frame: During tDCS or sham stimulation. Day 1 for non-smokers. Day 1 or 2 for smokers (counterbalanced for nicotine condition)
Measure: Mean (Standard Deviation); unit: 1/sec
Arm/Group | tDCS Arm - Non-smoker | tDCS Arm - Sated Smoker | tDCS Arm - Withdrawn Smoker
Number analyzed (Participants) | 28 | 15 | 15
1/sec
  Reaction speed - Anodal left dlPFC stimulation - shapes condition | 1.06 (.19) | 1.18 (.26) | 1.07 (.25)
  Reaction speed - Anodal left dlPFC stimulation - faces condition | .90 (.12) | 1.00 (.24) | .89 (.32)
  Reaction speed - Cathodal left dlPFC stimulation - shapes condition | 1.04 (.20) | 1.2 (.25) | 1.0 (.28)
  Reaction speed - Cathodal left dlPFC stimulation - faces condition | .93 (.18) | 1.0 (.27) | .82 (.27)
  Reaction speed - Sham stimulation - shapes condition | 1.02 (.18) | 1.22 (.27) | 1.05 (.27)
  Reaction speed - Sham stimulation - faces condition | .88 (.15) | 1.0 (.26) | .86 (.26)

9. Primary Outcome: Nicotine Withdrawal From WSWS
Description: Nicotine withdrawal as measured from the total score on the Wisconsin Smoking Withdrawal Scale (WSWS). The WSWS is a 28-item questionnaire ranging from 0 (strongly disagree) to 4 (strongly agree). The total score ranges from 0 to 112, with higher scores indicating more withdrawal symptoms. Cigarette smokers were 12 hour (overnight) abstinent and had either a nicotine patch or a placebo patch placed 1-2 hours before scanning.
Time Frame: 12 hours nicotine abstinent (plus 1-2 hours after patch)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Main Arm - Sated Smoker | Main Arm - Withdrawn Smoker
Number analyzed (Participants) | 30 | 30
score on a scale | 43.5 (2.6) | 50.8 (3.1)

10. Primary Outcome: Nicotine Craving From TCQ-SF
Description: Nicotine craving as measured from the total score on the Tobacco Craving Questionnaire-Short Form (TCQ-SF). The TCQ-SF is a 12-item questionnaire designed to measure craving for cigarettes. Each question is answered on a 7-point scale from 1 (Strongly Disagree) to 7 (Strongly Agree). Total scores range from 12 to 84, with higher scores indicating more craving.
  Cigarette smokers were 12 hour (overnight) abstinent and had either a nicotine patch or a placebo patch placed 1-2 hours before scanning.
Time Frame: 12 hours nicotine abstinent (plus 1-2 hours after patch)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Main Arm - Sated Smoker | Main Arm - Withdrawn Smoker
Number analyzed (Participants) | 30 | 30
score on a scale | 46.7 (2.9) | 51.9 (3.6)

11. Primary Outcome: Affect From PANAS
Description: Positive and Negative mood from the Positive and Negative Affect Schedule (PANAS). The PANAS consists of 20 words related to emotions that participants indicate to what extent they felt this way in the last week. Words are rated from 1 (very slightly or not at all) to 5 (extremely). The PANAS is broken into a Positive and Negative subscale, each consisting of 10 questions and thus ranging from 10 to 50. Higher numbers are indicative of higher levels of positive affect and higher levels of negative affect respectively.
  Cigarette smokers were 12 hour (overnight) abstinent, and had either a nicotine patch or a placebo patch placed 1-2 hours before scanning.
Time Frame: 12 hours nicotine abstinent (plus 1-2 hours after patch)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Main Arm - Sated Smoker | Main Arm - Withdrawn Smoker
Number analyzed (Participants) | 30 | 30
score on a scale
  Positive Subscale | 34.8 (1.4) | 31.2 (1.3)
  Negative Subscale | 11.7 (0.4) | 13.3 (1.0)

ADVERSE EVENTS:
Time Frame: From baseline to Scan 2 for tDCS Smoker arm (including behavioral pilot). Approximately 1 week to 3 months total. From Scan 1 to Scan 2 for tDCS non-smoker arm (including behavioral pilot). Approximately 1 week to 3 months total. From Phase 1 (pre-treatment study visits) to Phase 3 (follow-up visits) for Treatment arm. Approximately 1 - 1.5 years total. Phase 1 only for non-treatment arm. Approximately 3 - 5 weeks total.
Groups:
- tDCS Arm - Non-Smoker; tDCS Arm - Behavioral Pilot: Healthy non-smoking, non-drug dependent controls
Arm/Group | Main Study - Treatment | Main Study - Non-Treatment | Main Study - Motivational Interviewing Arm | tDCS Arm - Smoker | tDCS Arm - Non-Smoker | tDCS Arm - Behavioral Pilot
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/28 | 0/2 | 0/32 | 0/33 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/28 | 0/2 | 0/32 | 0/33 | 0/3
Other Adverse Events (participants affected / at risk) | 0/14 | 5/28 | 0/2 | 7/32 | 3/33 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study - Treatment (N=14) | Main Study - Non-Treatment (N=28) | Main Study - Motivational Interviewing Arm (N=2) | tDCS Arm - Smoker (N=32) | tDCS Arm - Non-Smoker (N=33) | tDCS Arm - Behavioral Pilot (N=3)
Headache (General disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Lower back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Elevated Blood Pressure (Cardiac disorders) | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shortness of Breath/Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Brief Psychotic Reaction (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Paranoia
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
General Warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — One particular participant reported an uncomfortable warm feeling in neck during tDCS in scanner.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT01511614/Prot_SAP_000.pdf